CLINICAL TRIAL: NCT06211400
Title: Vibration Exercise for Crohn's to Observe Response
Acronym: VECTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Collaborators: University of Central Lancashire (Other); Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VECTOR
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration Exercise (Experimental)
  Interventions: Other: Whole body vibration exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Whole body vibration exercise — 6-week supervised whole body vibration exercise programme (training sessions three times per week lasting 10 min) alongside a lifestyle education programme
  Arms: Vibration Exercise

SUMMARY:
Background: Crohn's disease (CD) is a long-term inflammatory condition of the digestive system. People with CD often have unpredictable and debilitating symptoms, including abdominal pain, diarrhoea and fatigue. In addition, they require long-term treatment with frequent negative effects and often need surgery and hospitalisations. Therefore, people with CD report a lower health-related quality of life (HRQOL) compared with other people. Doctors are constantly trying to find new treatments to improve HRQOL and control symptoms and whole body vibration exercise could be a potential treatment.

Exercise might be a simple, safe, and low-cost intervention for improving HRQOL in people with CD. This is because it has the potential to improve several aspects of physical, mental and social well-being simultaneously. Adults with CD have been shown to be less active than the general population and do not meet the recommended daily physical activity guidelines. One barrier to exercise is lack of time, however whole-body vibration exercise (where you stand and squat on a vibrating plate) can be done over a much shorter duration and at a lower intensity to gain potentially similar or at times greater benefits. More research is needed to understand the effects, both positive and negative of vibration exercise in people with CD.

Aim: This study begins to understand whether undertaking a supervised 6-week vibration exercise programme for adults with mild to moderately active Crohn's disease improves HRQoL and other symptoms such as fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18-65 years old
* Clinical diagnosis of CD for at least 4 weeks before randomization

  * Mild to moderate active CD (150-220 CDAI)
  * Stable medication for at least 4 weeks before randomization
  * Able to provide written consent, complete the study questionnaires and travel to the research centre for study assessment visits and exercise sessions
  * Be doing less than 60 minutes of purposeful exercise per week

Exclusion Criteria:

* Over 65 years old Severe or uncontrolled medical conditions that make it undesirable for the patient to participate

  * Coexistent serious autoimmune disease such as rheumatoid arthritis or systemic sclerosis
  * Planned major surgery within the first 3 months after randomization
  * Are pregnant, or are planning pregnancy within the first 3 months after randomization
  * Poor tolerability to venepuncture or lack of adequate venous access for required blood sampling
  * Current participation in >60 min/week of purposeful exercise, such as jogging or cycling
  * Participation in another clinical trial for which concurrent participation is deemed inappropriate
  * Any orthopaedic implants (hip, knee, spine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | change in IBDQ from baseline to 6 weeks
  The scale has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health).

SECONDARY OUTCOMES:
Crohn's disease activity index (CDAI) | change in CDAI from baseline to 6 weeks
  CDAI is a clinically assessed measure of disease activity in Crohn's patients. The score ranges from 0-600 with higher scores being indicative of higher disease activity
Concentration of Faecal Calprotectin (FC) | change in FC from baseline to 6 weeks
  a marker of inflammation in the gastrointestinal tract. Higher levels are indicative of higher inflammation levels
Inflammatory Bowel Disease Fatigue (IBD Fatigue) | change in IBD fatigue from baseline to 6 weeks
  The IBD Fatigue Scale is comprised of two components. Part 1 the questionnaire will identify fatigue, its severity, frequency and duration and scores range from 0-20 with a higher score meaning greater fatigue. Part 2 assesses the perceived impact of fatigue on your daily activities and scores range from 0-120 with a higher score meaning greater perceived impact.
Hospital Anxiety and Depression (HADS) | change in HADS from baseline to 6 weeks
  The Hospital Anxiety and Depression Scale measures anxiety and depression in patients. A higher score indicates greater anxiety and depression.
Perceived pain | change in pain from baseline to 6 weeks
  visual analogue scale from 0-10, 0 being no pain and 10 being most intense pain possible
Estimated Cardiorespiratory fitness | change in estimated maximal oxygen consumption from baseline to 6 weeks
  Chester step test to estimate maximal oxygen consumption. It involves stepping in time to a metronome and measuring heart rate.
Concentration of Tnf-alpha | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Interleukin-6 (IL6) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Interleuken-10 (IL10) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Interleukin 17a (IL17a) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Interleukin 12 (IL12) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Interleukin 23 (IL23) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation
Concentration of Transforming Growth Factor Beta (TGF-Beta) | change from baseline to 6 weeks
  This measure will be obtained from blood samples to provide a measure of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hertfordshire, Hatfield, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No